CLINICAL TRIAL: NCT06063538
Title: A Prospective Study Using Intra-Pericardial Amiodarone for the Prevention of Postoperative Atrial Fibrillation (POAF) in Patients Undergoing Cardiac Arterial Bypass Grafting and/or Valve Surgery
Brief Title: Prevention of Postoperative Atrial Fibrillation (POAF) Using Intra-Pericardial Amiodarone
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Helios Cardio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-0847
Record Dates: First submitted 2023-09-21; First posted 2023-10-02 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation; Post-Op Complication
MeSH Terms: conditions — Atrial Fibrillation; Postoperative Complications | interventions — Amiodarone

STUDY DESIGN:
Intervention Model Description: To demonstrate that there is no systemic presence of amiodarone, the first three patient will receive 600 mg amiodarone into the intact pericardial space (IPS). Amiodarone serum levels will be tested at post operative days 2 and 6. The study will only proceed if there is a serum amiodarone level less than 25% of the normal therapeutic level. This should insure lack of systemic toxicity. After the first 3 patients have demonstrated low amiodarone blood levels, a total of up to 60 patients will be enrolled in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CardiaMend Pericardial and Epicardial Reconstruction Matrix used in combination with amiodarone (Experimental): Patients randomized to this study arm includes the CardiaMend which will be used according to the instructions for use. It will be patted dry to facilitate implantation. Pieces will be cut to cover the right and left atria. The remaining piece will be contoured to close the anterior pericardial space. Four ampules of amiodarone (150mg/3ml; 12cc total volume) will be drawn into a syringe. 2cc will be dripped over the right atrium and a small CardiaMend patch placed to cover this area. Another 2cc will be used over the left atrium and covered with the CardiaMend. The anterior pericardial space will be closed without putting pressure on the underlying structures using the CardiaMend attached to the native pericardium utilizing running 4-0 monofilament suture.
  Interventions: Combination Product: CardiaMend in Combination with Amiodarone
- University of Chicago's standard of care in patients undergoing isolated CABG or valve surgery (No Intervention): The standard of care for this study at The University of Chicago is to ligate the left atrial appendage (LAA) during the proposed cardiac surgery (intra-operative) to reduce the occurrence of post operative atrial fibrillation (A-FIB) in combination with amiodarone injections (if applicable).

INTERVENTIONS:
Combination Product: CardiaMend in Combination with Amiodarone — The first three patient will receive 600 mg amiodarone into the intact pericardial space. Amiodarone serum levels will be tested at post operative days 2 and 6. The study will only proceed if there is a serum amiodarone level less than 25% of the normal therapeutic level. This should insure lack of systemic toxicity. After the first 3 patients have demonstrated low amiodarone blood levels, a total of up to 60 patients will be enrolled in the study.
  The CardiaMend patch will saturated per the instructions and be sutured into place. Amiodarone will be dripped directly over the heart.
  Arms: CardiaMend Pericardial and Epicardial Reconstruction Matrix used in combination with amiodarone

SUMMARY:
The purpose of this study is to evaluate the combination of CardiaMend, with the addition of amiodarone in the prevention of postoperative atrial fibrillation (POAF) in patients undergoing cardiac arterial bypass grafting (CABG) or valve surgery.

DETAILED DESCRIPTION:
This study involves using CardiaMend, an FDA cleared (K210331) pericardial reconstruction matrix with the addition of amiodarone, an FDA approved antiarrhythmic drug, as a prevention of post operative atrial fibrillation.

This is a single-center, prospective randomized study enrolling adult subjects undergoing isolated cardiac arterial bypass or valve surgery, via complete median sternotomy.

CardiaMend will be used according to the Instructions for Use, and then patted dry to facilitate implantation. Four ampules of amiodarone (150mg/3ml; 12cc total volume) will be drawn into a syringe. 2cc will be dripped over the right atrium and a small CardiaMend patch placed to cover this area. Another 2cc will be used over the left atrium and covered with the CardiaMend. The anterior pericardial space will be closed without putting pressure on the underlying structures using the CardiaMend attached to the native pericardium utilizing running 4-0 monofilament suture. A small edge may be left open for drain placement and a small slit for the Left Internal Mammary Artery (LIMA) in case of CABG. The remaining 8 cc of amiodarone will be instilled to the closed pericardial space.

Patients will have continuous electrocardiogram (EKG) until discharge. If clinically indicated, patients will receive a monitor for home monitoring per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 20-85 years old.
* Patients able to provide written informed consent, understand, and be willing to comply with study-related procedures.
* Participants who are scheduled to undergo open-chest cardiac surgery via complete median sternotomy. Includes:

  * Coronary artery bypass graft (CABG) and/or valve repair/replacement procedures (aortic, mitral, or tricuspid)
  * Isolated ascending aortic aneurysm replacement/repair
  * Note: Left atrial appendage (LAA) procedures are allowed if CABG and/or valve repair or replacement is the qualifying surgical procedure, but is not a qualifying surgical procedure on its own.
* In sinus rhythm at the time of office visit and prior electrocardiogram (EKG) (note: continuous EKG monitoring for 48 hours is not required).

Exclusion Criteria:

* Subject unable to give voluntary written informed consent, is unlikely to cooperate or is legally incompetent, including subjects who are institutionalized by court or official order, or in a dependency relationship with, testing center or investigator.
* Any condition which could interfere with the subject's ability to comply with the study.
* Ongoing participation in an interventional clinical study or during the preceding 30 days.
* Female subjects who are pregnant, breastfeeding, were pregnant within the last three months, or are planning to become pregnant during the course of the study.
* Active skin or deep infection at the site of implantation.
* History of chronic wounds or wound-healing disorders.
* Known connective tissue diseases (e.g. Ehlers-Danlos syndrome, Epidermolysis bullosa, Marfan syndrome, Osteogenesis imperfecta).
* Immune-suppressed subjects, immune-deficiency subjects (properly managed diabetes mellitus is not an exclusion criterion).
* Concomitant oral or IV systemic corticosteroid therapy and/or other constant anti-inflammatory therapies.
* Patients already receiving amiodarone as a treatment for atrial fibrillation or ventricular arrhythmias.
* Disease of the left pleura, previous intervention in the left pleural space, or chest deformity.
* Subjects with end-stage chronic-renal disease / dialysis.
* STS (Society of Thoracic Surgeons Score) risk score >5.5% for 30 day mortality.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Post Operative Atrial Fibrillation | Through discharge, an average 7 days to 2 weeks
  The patients have continuous electrocardiogram (EKG) monitoring until discharge to evaluate for any evidence of atrial fibrillation or atrial flutter which lasts longer than one hour or if less than one hour, requires medical or procedural intervention. Evidence of atrial fibrillation or atrial flutter will be confirmed by 12 lead electrocardiogram by loss or changes to the P wave, as well as irregularities in the QRS wave interval, heart rhythm, or rate. If clinically indicated, patients will receive a monitor for home monitoring per standard of care.

SECONDARY OUTCOMES:
Additional Hospital Time Required Due to Atrial Fibrillation/Flutter | Through discharge, an average 7 days to 2 weeks
  Burden of atrial fibrillation as defined by additional treatment regimen, additional time in intensive care unit (ICU), complications directly associated with atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Valluvan Jeevanandam, MD, Principal Investigator — Director of Heart and Vascular Center
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Helios Cardio Inc., who will be the study collaborator will have access to only de-identified form of the data.

REFERENCES:
- [Background] Habbab LM, Chu FV. Intrapericardial Amiodarone for the Prevention of Postoperative Atrial Fibrillation. J Card Surg. 2016 Apr;31(4):253-8. doi: 10.1111/jocs.12700. Epub 2016 Feb 2. PMID 26833498
- [Background] Camm AJ. Safety considerations in the pharmacological management of atrial fibrillation. Int J Cardiol. 2008 Jul 21;127(3):299-306. doi: 10.1016/j.ijcard.2007.11.006. Epub 2008 Jan 8. PMID 18191470
- [Background] Frendl G, Sodickson AC, Chung MK, Waldo AL, Gersh BJ, Tisdale JE, Calkins H, Aranki S, Kaneko T, Cassivi S, Smith SC Jr, Darbar D, Wee JO, Waddell TK, Amar D, Adler D; American Association for Thoracic Surgery. 2014 AATS guidelines for the prevention and management of perioperative atrial fibrillation and flutter for thoracic surgical procedures. J Thorac Cardiovasc Surg. 2014 Sep;148(3):e153-93. doi: 10.1016/j.jtcvs.2014.06.036. Epub 2014 Jun 30. No abstract available. PMID 25129609
- [Background] Beau J, Kulik A. Topical amiodarone to prevent postoperative atrial fibrillation: Need for further study. J Thorac Cardiovasc Surg. 2016 Feb;151(2):600. doi: 10.1016/j.jtcvs.2015.10.007. No abstract available. PMID 26806512
- [Background] de Lima Conceicao MR, Teixeira-Fonseca JL, Marques LP, Souza DS, da Silva Alcantara F, Orts DJB, Roman-Campos D. Extracellular acidification reveals the antiarrhythmic properties of amiodarone related to late sodium current-induced atrial arrhythmia. Pharmacol Rep. 2024 Jun;76(3):585-599. doi: 10.1007/s43440-024-00597-2. Epub 2024 Apr 15. PMID 38619735
- [Background] Egan S, Collins-Smyth C, Chitnis S, Head J, Chiu A, Bhatti G, McLean SR. Prevention of postoperative atrial fibrillation in cardiac surgery: a quality improvement project. Can J Anaesth. 2023 Dec;70(12):1880-1891. doi: 10.1007/s12630-023-02619-8. Epub 2023 Nov 2. PMID 37919634
- [Background] Piccini JP, Ahlsson A, Dorian P, Gillinov AM, Kowey PR, Mack MJ, Milano CA, Noiseux N, Perrault LP, Ryan W, Steinberg JS, Voisine P, Waldron NH, Gleason KJ, Titanji W, Leaback RD, O'Sullivan A, Ferguson WG, Benussi S; NOVA-AF Investigators. Efficacy and Safety of Botulinum Toxin Type A for the Prevention of Postoperative Atrial Fibrillation. JACC Clin Electrophysiol. 2024 May;10(5):930-940. doi: 10.1016/j.jacep.2024.01.020. Epub 2024 Apr 24. PMID 38661602
- [Result] Echahidi N, Pibarot P, O'Hara G, Mathieu P. Mechanisms, prevention, and treatment of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Feb 26;51(8):793-801. doi: 10.1016/j.jacc.2007.10.043. PMID 18294562
- [Result] Lowres N, Mulcahy G, Jin K, Gallagher R, Neubeck L, Freedman B. Incidence of postoperative atrial fibrillation recurrence in patients discharged in sinus rhythm after cardiac surgery: a systematic review and meta-analysis. Interact Cardiovasc Thorac Surg. 2018 Mar 1;26(3):504-511. doi: 10.1093/icvts/ivx348. PMID 29161419
- [Result] Rego A, Cheung PC, Harris WJ, Brady KM, Newman J, Still R. Pericardial closure with extracellular matrix scaffold following cardiac surgery associated with a reduction of postoperative complications and 30-day hospital readmissions. J Cardiothorac Surg. 2019 Mar 15;14(1):61. doi: 10.1186/s13019-019-0871-5. PMID 30876459
- [Result] Feng XD, Wang XN, Yuan XH, Wang W. Effectiveness of biatrial epicardial application of amiodarone-releasing adhesive hydrogel to prevent postoperative atrial fibrillation. J Thorac Cardiovasc Surg. 2014 Sep;148(3):939-43. doi: 10.1016/j.jtcvs.2014.05.049. Epub 2014 May 22. PMID 25043862
- [Result] Ayers GM, Rho TH, Ben-David J, Besch HR Jr, Zipes DP. Amiodarone instilled into the canine pericardial sac migrates transmurally to produce electrophysiologic effects and suppress atrial fibrillation. J Cardiovasc Electrophysiol. 1996 Aug;7(8):713-21. doi: 10.1111/j.1540-8167.1996.tb00579.x. PMID 8856462
- [Result] Darsinos JT, Karli JN, Samouilidou EC, Krumbholz B, Pistevos AC, Levis GM. Distribution of amiodarone in heart tissues following intrapericardial administration. Int J Clin Pharmacol Ther. 1999 Jun;37(6):301-6. PMID 10395122
- [Result] Marcano J, Campos K, Rodriguez V, Handy K, Brewer MA, Cohn WE. Intrapericardial delivery of amiodarone rapidly achieves therapeutic levels in the atrium. Heart Surg Forum. 2013 Oct;16(5):E279-86. doi: 10.1532/hsf98.2013188. PMID 24364084